CLINICAL TRIAL: NCT04232241
Title: Matched Unrelated vs. Haploidentical Donor for Allogeneic Stem Cell Transplantation in Patients With Acute Leukemia With Identical GVHD Prophylaxis - A Randomized Prospective European Trial.
Brief Title: Matched Unrelated vs. Haploidentical Donor for Allogeneic Stem Cell Transplantation in Patients With Acute Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: GKM Gesellschaft für Therapieforschung mbH (Unknown); Staburo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HaploMUDStudy
Record Dates: First submitted 2020-01-02; First posted 2020-01-18 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia in Remission; Acute Lymphoblastic Leukemia in Remission; Myelodysplastic Syndromes
Keywords: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Allogeneic Stem Cell Transplantation; Matched Unrelated Allogeneic Stem Cell Transplantation; Haploidentical Allogeneic Stem Cell Transplantation; anti-leukemic activity; Cyclophosphamide as GVHD prophylaxis
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (Active Comparator): Allogeneic stem cell transplantation from 10/10 HLA matched unrelated donor
  Interventions: Drug: Allogeneic Stem Cell Transplantation
- Treatment B (Experimental): Allogeneic stem cell transplantation from haploidentical donor
  Interventions: Drug: Allogeneic Stem Cell Transplantation

INTERVENTIONS:
Drug: Allogeneic Stem Cell Transplantation — Allogeneic Stem Cell Transplantation

SUMMARY:
Primary objective of this open label, two-arm, multicenter, multinational, randomized trial is to compare anti-leukemic activity of allogeneic stem cell transplantation for patients with acute leukemia in complete remission between a 10/10 HLA matched unrelated donor and a haploidentical donor.

The hypothesis: Haploidentical stem cell transplantation with post cyclophosphamide induces a stronger anti-leukemic activity in comparison to 10/10 HLA matched unrelated donor and reduces the risk of relapse at 2 years after stem cell transplantation by 10%.

DETAILED DESCRIPTION:
Secondary objectives are to assess and compare the safety and efficacy of study treatments therapy in both study arms on non-relapse mortality (NRM), relapse-free survival (RFS), Overall survival (OS), QOL, toxicity, development of acute and chronic GvDH as well as engraftment and chimerism and impact of measurable residual disease.

ELIGIBILITY:
Inclusion Criteria

1. Acute Myeloid Leukemia (AML) intermediate or high risk according to ELN or Acute Lymphoblastic Leukemia (ALL) high risk according to ESMO guidelines in 1. CR or AML/ALL in 2. CR, or high risk MDS (according to IPSS-R) in 1. CR or 2. CR.
2. Patients age: 18 - 70 years at time of inclusion (female and male).
3. Patients understand and voluntarily sign an informed consent form.
4. ECOG ≤ 2.
5. 10/10 HLA-matched unrelated donor and haploidentical (≥ 5/10 and ≤ 8/10 HLA) relative matched donor available at least 4 weeks after completion of induction and/or consolidation therapy.
6. Females/Males who agree to comply with the applicable contraceptive requirements of the protocol.

Exclusion Criteria

1. Severe renal, hepatic, pulmonary or cardiac disease, such as:

   * total bilirubin, SGPT or SGOT > 3 times upper the normal level
   * left ventricular ejection fraction < 30 %
   * creatinine clearance < 30 ml/min
   * DLCO < 35 % and/or receiving supplementary continuous oxygen
2. Positive serology for HIV.
3. Pregnant or lactating women (positive serum pregnancy test).
4. Age < 18 and ≥ 71 years.
5. Uncontrolled invasive fungal infection at time of screening (baseline).
6. Serious psychiatric or psychological disorders.
7. Participation in another study with ongoing use of unlicensed investigational product from 28 days before study enrollment.
8. Uncontrolled severe autoimmune disease or uncontrolled other malignancy.
9. Availability of an HLA-identical sibling as donor source.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Relapse incidence at two years between both arms | 2 years
  The primary efficacy endpoint will be analyzed using cumulative incidence estimation to assess the subdistribution hazard rates for both treatment groups at two years after accounting for competing risk events.

SECONDARY OUTCOMES:
Overall survival at two years between both arms | 2 years
  The overall survival at two years between both arms will be presented with Kaplan-Meier's estimates of survival.
Overall survival for all patients assigned to one of the two treatment arms as time to event endpoint | through study completion, an average of two yeras
  The overall survival for all patients will be presented with Kaplan-Meier curve. To compare the survival distributions between two arms, log-rank test will be performed, and two-sided p-values will be presented.
  If applicable, Cox regression model stratified by the types of leukemia, types of complete remission and conditioning will be performed as sensitivity analysis.
Comparison of GVHD/relapse-free survival as Composite endpoint in both arms | Starting at day +30 (+/- 3 d) to 24 months (+/- 1 mo) after allogenic stem cell transplantation (SCT)
  The rate of composite endpoint in both arms will be analyzed with the same methods as for the overall survival at two years between both arms.
Comparison of non-relapsed mortality (NRM) at 1 and 2 years after allogeneic SCT in both arms | At 1 and 2 years after allogeneic SCT
  Due to the existence of competing risk events (persisting disease and relapse), NRM of each arm at 1 and 2 years after allogeneic SCT will be analyzed with the same methods as for the primary endpoint
Comparison of acute graft-versus-host disease (aGVHD) on day +100 and 1 year (max grade) after allogeneic SCT according to the Glucksberg scale revised by Przepiorka et al. between both arms | On day +100 and 1 year (max grade) after allogeneic SCT
  For each time point, the frequency and percentage of aGVHD (maximum grade) of each arm will be presented. To compare the difference between both arms, logistic regression adjusted for covariates and stratification factors will be performed.
Comparison of chronic graft-versus-host disease (cGVHD) according to the NIH consensus criteria of Jagasia et al. at 1 and 2 years after allogeneic SCT between both arms | At 1 and 2 years after allogeneic SCT
  For each time point, the frequency and percentage of cGVHD of each arm will be presented. To compare the difference between both arms, logistic regression adjusted for the stratification factors will be performed.
Comparison of toxicity of both regimens scored according to the current version of the NCI CTCAE between both arms | through study completion, an average of two yeras
  Safety will be analyzed with frequency of patients with AEs as described above.
Comparison of immune reconstitution between both arms | At day 30, 100, 6 months, 1 year and 2 years after allogenic SCT
  Frequency and percentage of patients having immune reconstitution in two arms will be provided. For the comparison between two arms, logistic regression adjusted for the stratification factors will be performed.
Comparison of full donor chimerism between both arms | At day 30, 100, 6 months, 1 year and 2 years after allogenic SCT
  Frequency and percentage of patients having full donor chimerism in two arms will be provided. For the comparison between two arms, logistic regression adjusted for the stratification factors will be performed.
Evaluation of Sorror Risk Score on outcome after allogeneic SCT | At baseline
  Comorbidity score after Sorror will be assessed prior to randomization and outcome in both arms will be analyzed according the pre-transplant Sorror score.
Comparison of QOL (FACT-BMT) before and after transplantation at + 100 days, 6 months, 1 year, 2 years between both arms | At day 100, 6 months, 1 year and 2 years after allogenic SCT
  The means of change in scores at each time point (day 100, 6 months, 1 year and 2 years after transplantation respectively) from baseline and the confidence intervals of each arm will be presented. To compare the difference in QOL scores between both arms, logistic regression adjusted for covariates and stratification factors will be performed for each time point.

OTHER OUTCOMES:
Scientific Endpoint (optional) | 2 years
  Comparison of relapse incidence at two years between MRD positive and negative patients in both arms
Scientific Endpoint (optional) | 2 years
  Comparison of overall survival at two years between MRD positive and negative patients in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kröger, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Stem Cell Transplantation
Locations (24):
- Austria (3):
  - LKH-Univ. Klinikum Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Medizinische Universität Wien, Universitätsklinik für Innere Medizin I Einrichtung für Stammzelltransplantation KMT, Vienna
- Institute of Hematology and Blood Transfusion, Prague, Czechia
- Turku University Central Hospital, Turku, Finland
- Germany (9):
  - University Hospital Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt am Main | Medizinische Klinik II, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Leipzig Dep. Innere Medizin, Neurologie und Dermatologie Medizinische Klinik und Poliklinik I - Hämatologie und Zelltherapie, Hämostaseologie, Leipzig
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
- ASST Papa Giovanni XXIII, Bergamo, Italy
- Pavlov First Saint Petersburg State Medical University, Saint Petersburg, Russia
- Spain (8):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanz J, Galimard JE, Labopin M, Afanasyev B, Sergeevich MI, Angelucci E, Kroger N, Koc Y, Ciceri F, Diez-Martin JL, Arat M, Sica S, Rovira M, Aljurf M, Tischer J, Savani B, Ruggeri A, Nagler A, Mohty M. Post-transplant cyclophosphamide containing regimens after matched sibling, matched unrelated and haploidentical donor transplants in patients with acute lymphoblastic leukemia in first complete remission, a comparative study of the ALWP of the EBMT. J Hematol Oncol. 2021 May 28;14(1):84. doi: 10.1186/s13045-021-01094-2. PMID 34049582